CLINICAL TRIAL: NCT02984579
Title: Multi-center Study to Assess the Non-inferiority of YD REBA MTB-MDR® and Hain GenoType® MTBDRplus V2 Line Probe Assays Compared to Hain GenoType® MTBDRplus V1
Brief Title: Line Probe Assay Evaluation Study
Acronym: YD
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Research Center Borstel (Other); National Institute for Communicable Diseases, South Africa (Other); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: YD7012-03
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Multidrug-Resistant Tuberculosis; Isoniazid Resistant Pulmonary Tuberculosis; Rifampicin Resistant Tuberculosis; Pulmonary Tuberculoses
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects: All strains in Phase 1 and all Sputum samples in Phase 2 were tested with Hain Genotype MTBDRplus V1, Hain Genotype MTBDRplus V2, and YD REBA MTB-MDR diagnostic tests.
  Investigators and Operators were blinded to all other results for a sample upon data entry.
  Interventions: Device: YD REBA MTB-MDR; Device: Hain Genotype MTBDRplus V1; Device: Hain Genotype MTBDRplus V2

INTERVENTIONS:
Device: YD REBA MTB-MDR — Conducted on stored, de-identified leftover samples. A line probe assay designed for detection of Multidrug-resistant tuberculosis (MDR-TB). The REBA MTB-MDR® assay is a qualitative in vitro test for the identification of Mycobacterium tuberculosis (MTB) complex and its susceptibility to rifampin and isoniazid from cultured samples and smear positive specimens.
Device: Hain Genotype MTBDRplus V1 — Conducted on stored, de-identified leftover samples. There is only one Line Probe Assay for molecular MTB drug resistance globally available, the GenoType® MTBDRplus V.1 from Hain Lifescience. This assay includes rpoB gene probes for Rifampin (RIF) resistance, katG gene probes for high level Isoniazid (INH) resistance, and inhA gene probes for determination of low level INH resistance
Device: Hain Genotype MTBDRplus V2 — Conducted on stored, de-identified leftover samples. An updated version of the Hain Genotype MTBDRplus V1 assay, the Genotype MTBDRplus V.2 line probe assay, showed increased sensitivity for MTB detection in the 2 studies published so far

SUMMARY:
This is a multi-center, blinded study to determine the performance of the YD Diagnostic Corporation (YD) REBA MTB-MDR® and Hain Genotype MTBDRplus V2 kit in a total of 600 clinical isolates and 900 residual sputum samples from patients with symptoms of pulmonary TB (PTB) and at risk of drug resistance. All testing was done on stored, de-identified leftover samples.

The study involved three World Health Organization (WHO) Supranational Reference Laboratories with well-characterized strain collections and access to sputum samples with significant rates of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Informed consent
* Patients evaluated for pulmonary TB

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consisted of two phases. In phase 1, each site was sent a different set of 200 clinical isolates from the Research and Training in Tropical Diseases and Institute for Tropical Medicine collections (ITM).
  In phase 2, samples from 274 patients recruited between Azerbaijan and Moldova were tested in Germany, while samples from 214 (locally-recruited) patients were tested in South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
INH/RIF Resistance Detection | At the end of study 9-10 Months after the Study started

SECONDARY OUTCOMES:
Multi-Drug Resistant TB detection | At the end of study 9-10 Months after the Study started
  Is the subject resistant to both INH and RIF